CLINICAL TRIAL: NCT04904770
Title: Time Performance of Scoop Stretcher Versus Vacuum Mattress for Prehospital Spinal Stabilization: Open-Label Simulation-based Randomized Controlled Trial
Brief Title: Time Performance of Scoop Stretcher Versus Vacuum Mattress for Prehospital Spinal Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneve TEAM Ambulances (Other)
Responsible Party: Principal Investigator, Stuby Loric, Principal Investigator, Geneve TEAM Ambulances
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSSS
Record Dates: First submitted 2021-05-16; First posted 2021-05-27 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Immobilization
Keywords: Spinal stabilization; Prehospital; Emergency Medical Services; Scoop stretcher; Vacuum mattress; Spinal cord injury; Prehospital emergency care
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Due to nature of therapy, it is impossible to mask participants, care provider, investigators or outcomes assessors. Statistician will however be blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scoop stretcher (Experimental): A scoop stretcher will be used as device to perform spinal stabilization
  Interventions: Device: Scoop stretcher
- Vacuum mattress (Active Comparator): A vacuum mattress will be used as device to perform spinal stabilization
  Interventions: Device: Vacuum mattress

INTERVENTIONS:
Device: Scoop stretcher — Already included in arm/group description
  Arms: Scoop stretcher
Device: Vacuum mattress — Already included in arm/group description
  Arms: Vacuum mattress

SUMMARY:
A simulation-based randomized controlled trial was designed with the objective to assess the time needed to achieve spinal stabilization using a scoop stretcher compared to a vacuum mattress.

DETAILED DESCRIPTION:
A simulation-based randomized controlled trial was designed with the objective to assess the time needed to achieve spinal stabilization using a scoop stretcher compared to a vacuum mattress. The participants will be recruited among healthcare workers from one Emergency Medical Service. Then, the participants will first act as patient and undergo spinal stabilization from an other team, afterwards they will have to complete a spinal stabilization either using a scoop stretcher or a vacuum mattress, depending on allocation regarding randomization. The sessions will be video recorded to allow subsequent assessment.

ELIGIBILITY:
Inclusion Criteria:

* registered paramedics or emergency medical technician (EMT) actually working in the ambulance service.

Exclusion Criteria:

* member of study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in time to perform the procedure | At study session (real-time assessment), in July or August
  The time required to complete the procedure from the team leader's order to start, until the device is left up from the ground, measured in seconds.

SECONDARY OUTCOMES:
Quality of stabilization | At study session (real-time assessment), in July or August
  Quality of stabilization (accuracy of tightening of restraints belts) regarding the standard operating procedure
Level of anxiety | 5 minutes after spinal stabilization, on a questionnaire
  Participants will estimate their level of anxiety on a visual analog scale from 0 = "No anxiety at all" to 10 = "The worst anxiety imaginable".
Level of comfort | 5 minutes after spinal stabilization, on a questionnaire
  Participants will estimate their level of comfort on a visual analog scale from 0 = "Very, very comfortable" to 10 = "Very, very uncomfortable".
Degree of induced dyspnoea or shortness of breath | 5 minutes after spinal stabilization, on a questionnaire
  Participants will estimate their degree of induced dyspnoea or shortness of breath on a visual analog scale from 0 = "No dyspnoea or shortness of breath" to 10 = "The worst imaginable dyspnoea".

CONTACTS AND LOCATIONS:
Overall Officials: Loric Stuby, Principal Investigator — Geneve TEAM Ambulances
Locations (1):
- Genève TEAM Ambulances, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Shared upon request
Supporting Information: ICF
Time Frame: Since publication, for 10 years
Access Criteria: Upon request